CLINICAL TRIAL: NCT03860909
Title: Assessment of Pelvic Endometriosis: Correlation of US and MRI With Laparoscopic Findings
Brief Title: Pelvic Endometriosis: Correlation of US and MRI With Laparoscopic Findings
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal yusef, principle investigator, Assiut University
Other Study IDs: AssiutU10
Record Dates: First submitted 2019-02-27; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometriosis is classically defined as the presence of endometrial glands and stroma outside the uterine cavity and its musculature.

The definition of deep endometriosis is based on anatomic assumptions that may prove erroneous.

In fact, the term '' deep endometriosis '' should be reserved for lesions in the retroperitoneal tissue. For practical purposes, several reports included in the so-called deep endometriosis the infiltrative forms that involve vital structures such as the bowel, ureters, and bladder, as well as forms such as many rectovaginal lesions. For the term ''deep'' to apply, there should be ectopic endometrial tissue penetrating the peritoneum more than 5 mm in depth.

The ectopic endometrium responds to hormonal stimulation with various degrees of cyclic hemorrhage which result in suggestive symptoms and appearances.

A common symptom is infertility. Pelvic pain is a frequent complaint among patients with endometriosis. Such pain generally manifests as secondary dysmenorrhea, worsening primary dysmenorrhea, dyspareunia, or even noncyclic lower abdominal pain and backaches. The pain may be site-specific when endometriosis is found in unusual locations outside the pelvis.

Diagnosis Physical examination and laparoscopic exploration may not allow diagnosis or prediction of the extension of deep pelvic endometriosis, especially in pelvic retroperitoneal sites.

Transvaginal sonography is recommended for diagnosis of endometriomas and endometriosis of the bladder but its value for assessment of superficial peritoneal lesions, ovarian foci, and deep pelvic endometriosis is uncertain.

MR imaging is now commonly used for diagnosis of endometriosis and provides a tremendous advantage over other methods of investigation, owing to the possibility of making a complete survey of the anterior and posterior compartments of the pelvis at one time.

MRI is becoming a mainstay of preoperative diagnosis, in particular for diagnosis deep infiltrating endometriosis.

DETAILED DESCRIPTION:
A prospective study including 30 Female patients of reproductive who were previously clinically diagnosed to have endometriotic lesions. these will be sent to our department to identify the extent of the lesions and clarify the exact location for proper treatment.

All patients were evaluated with ultrasound and MRI. the sensitivity, specificity and diagnostic accuracy for both examination were calculated.

Transvaginal ultrasound and MRI will be done in our Radiology department to all patients after signing an informed consent to be enrolled in the study.

All our imaging results were finally compared to the laparoscopic results which are our gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who have symptoms consistent with endometriosis such as pelvic pain, dysmenorrhea, deep dyspareunia, and infertility

Exclusion Criteria:

* The common contraindication to MRI, peacemaker, metallic foreign bodies, and claustrophobia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: females with endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of Mri with Us in correlation with laparoscopic findings in female patients with endometriosis | one year
  comparison between MRI imaging and ultrasound combined with laproscopy in diagnosis of endometriosis

SECONDARY OUTCOMES:
The additive value of Mri in diagnosis of endometriosis | one year
  MRI better than ultrasound in diagnosis of endometriosis in correlated with laproscopy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abrao MS, Goncalves MO, Dias JA Jr, Podgaec S, Chamie LP, Blasbalg R. Comparison between clinical examination, transvaginal sonography and magnetic resonance imaging for the diagnosis of deep endometriosis. Hum Reprod. 2007 Dec;22(12):3092-7. doi: 10.1093/humrep/dem187. Epub 2007 Oct 18. PMID 17947378
- [Background] Anaf V, Simon P, El Nakadi I, Fayt I, Buxant F, Simonart T, Peny MO, Noel JC. Relationship between endometriotic foci and nerves in rectovaginal endometriotic nodules. Hum Reprod. 2000 Aug;15(8):1744-50. doi: 10.1093/humrep/15.8.1744. PMID 10920097
- [Background] Bazot M, Malzy P, Cortez A, Roseau G, Amouyal P, Darai E. Accuracy of transvaginal sonography and rectal endoscopic sonography in the diagnosis of deep infiltrating endometriosis. Ultrasound Obstet Gynecol. 2007 Dec;30(7):994-1001. doi: 10.1002/uog.4070. PMID 17992706
- [Background] Ros C, Martinez-Serrano MJ, Rius M, Abrao MS, Munros J, Martinez-Zamora MA, Gracia M, Carmona F. Bowel Preparation Improves the Accuracy of Transvaginal Ultrasound in the Diagnosis of Rectosigmoid Deep Infiltrating Endometriosis: A Prospective Study. J Minim Invasive Gynecol. 2017 Nov-Dec;24(7):1145-1151. doi: 10.1016/j.jmig.2017.06.024. Epub 2017 Jun 30. PMID 28673872
- [Background] Zhang JL. Functional Magnetic Resonance Imaging of the Kidneys-With and Without Gadolinium-Based Contrast. Adv Chronic Kidney Dis. 2017 May;24(3):162-168. doi: 10.1053/j.ackd.2017.03.006. PMID 28501079
- [Background] Whittaker CS, Coady A, Culver L, Rustin G, Padwick M, Padhani AR. Diffusion-weighted MR imaging of female pelvic tumors: a pictorial review. Radiographics. 2009 May-Jun;29(3):759-74; discussion 774-8. doi: 10.1148/rg.293085130. PMID 19448114
- [Background] Marcal L, Nothaft MA, Coelho F, Choi H. Deep pelvic endometriosis: MR imaging. Abdom Imaging. 2010 Dec;35(6):708-15. doi: 10.1007/s00261-010-9611-y. PMID 20390267
- [Background] Koninckx PR, Martin D. Treatment of deeply infiltrating endometriosis. Curr Opin Obstet Gynecol. 1994 Jun;6(3):231-41. PMID 8038409
- [Background] Mais V, Guerriero S, Ajossa S, Angiolucci M, Paoletti AM, Melis GB. The efficiency of transvaginal ultrasonography in the diagnosis of endometrioma. Fertil Steril. 1993 Nov;60(5):776-80. doi: 10.1016/s0015-0282(16)56275-x. PMID 8224260
- [Background] Guerriero S, Mais V, Ajossa S, Paoletti AM, Angiolucci M, Labate F, Melis GB. The role of endovaginal ultrasound in differentiating endometriomas from other ovarian cysts. Clin Exp Obstet Gynecol. 1995;22(1):20-2. PMID 7736636
- [Background] Fedele L, Bianchi S, Raffaelli R, Portuese A. Pre-operative assessment of bladder endometriosis. Hum Reprod. 1997 Nov;12(11):2519-22. doi: 10.1093/humrep/12.11.2519. PMID 9436698
- [Background] Roseau G, Dumontier I, Palazzo L, Chapron C, Dousset B, Chaussade S, Dubuisson JB, Couturier D. Rectosigmoid endometriosis: endoscopic ultrasound features and clinical implications. Endoscopy. 2000 Jul;32(7):525-30. doi: 10.1055/s-2000-9008. PMID 10917184